CLINICAL TRIAL: NCT03141502
Title: The New Skin Stretching Device for Treatment of Limb Tension Wounds: A Multicenter Randomized Controlled Clinical Study
Brief Title: The New Skin Stretching Device for Treatment of Limb Tension Wounds
Acronym: SSDRCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCSY2017-05
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-04

CONDITIONS: Trauma; Fractures, Open; Wounds and Injuries; Skin Expander
Keywords: tension wound; skin stretching device; skin grafting
MeSH Terms: conditions — Wounds and Injuries; Fractures, Open | interventions — Skin Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Stretching Device (SSD) (Experimental): the wound is primarily closed by aid of the SSD after necessary surgical debridement.
  Interventions: Device: Skin stretching device (SSD)
- Skin Grafting (SG) (Active Comparator): the wound is primarily closed by the technique of skin grafting after necessary surgical debridement.
  Interventions: Procedure: Skin grafting

INTERVENTIONS:
Device: Skin stretching device (SSD) — By making use of skin viscoelasticity, the special metal crochet of SSD would be embedded in both sides skin of the wound. Multiple cycles of stretching and relaxing wound lead to extended skin, changing the high tension incision into a low tension incision and facilitating the direct suture.
  Arms: Skin Stretching Device (SSD)
Procedure: Skin grafting — the standard technique of skin grafting after wound preparation.
  Arms: Skin Grafting (SG)

SUMMARY:
A randomized controlled trial is performed to evaluate the effectiveness and safety of the Skin Stretching Device (SSD) on limb tension incision closure by comparing whether the differences in wounds area, wounds closure time and scar assessment between the SSD and the skin grafting are statistically significant.

DETAILED DESCRIPTION:
Design:

This study is a multicenter and randomized control study with the participation of 15 major national or regional central hospitals. And the whole sample size is set to be 100 patients.

Patients who have been screened by inclusion and exclusion criteria will be randomly (non-transparent envelope) assigned to Skin Stretching Group (SS Group) or Skin Grafting Group (SG Group). Patients of both group will undergo surgical debridement for the same principle, while the Skin Stretching Device is used for the patients of SS Group for incision closure and the Skin Grafting is used for the patients of SG group for incision closure.

Outcome evaluation:

Wound and scar evaluation during surgery, three and six months after surgery will include the following parameters:

* surface area;
* Vancouver scar scale (VSS)
* vascularization and pigmentation;
* dermal architecture. After 3 and 6 months patients will undergo a biopsy of the scar under local anesthesia. The experimental group, treated with the SSD will undergo one extra biopsy of the formerly stretched skin.

Safety evaluation:

During the trial, adverse events are observed and evaluated. Adverse reactions to clinical manifestations are followed and recorded till the symptoms disappear. The subject with serious adverse events shall withdraw from the study and be treated accordingly.

ELIGIBILITY:
Inclusion criteria:

1. Age≥18 years old
2. Tension incision that cannot be directly closed due to limb trauma or surgical debridement
3. Incision that cannot be directly closed after the incision decompression for fascia compartment syndrome and ischemia and reperfusion injury
4. Both sides of the incision skin suitable for skin stretching

Exclusion criteria:

1. Age <18 years old
2. Skin disease
3. Keloid history
4. Local or systemic use of hormones
5. Systemic diseases: for example, diabetes, immunodeficiency disease, vascular disease and etc.
6. Other poor general state to result in inability for trial;
7. Mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-11 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
the change of surface area of the scar | change from surgery at 6 months
  it is performed by tracing the area of the scar directly onto non-stretchable transparent sterile sheets. then digitized and analyzed by software.

SECONDARY OUTCOMES:
Operation time | during surgery
  refers to the time required for the application of skin stretching device or skin grafting
Wound site and wound healing time | from surgery to 6 months
  record the site of the operation, and the time from the beginning of surgery to the complete healing of the wound.
Vancouver scar scale (VSS) | 3 and 6 months after surgery
  evaluate the scar scale by VSS
scar vascularization index | 3 and 6 months after surgery
  use photometric analyzer to measure its erythema index, assessing its angiogenesis and vascularization
scar pigmentation index | 3 and 6 months after surgery
  use photometric analyzer to measure its melanin index, assessing its pigmentation
collagen fibers arrangement under electron microscopy | surgery and 6 months after surgery
  use the drilling device to take the skin tissue of the diameter of 3mm for histological examination, measuring the collagen fibers arrangement by Electron microscopy
dermal matrix arrangement under electron microscopy | surgery and 6 months after surgery
  use the drilling device to take the skin tissue of the diameter of 3mm for histological examination, measuring the dermal matrix arrangement by Electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Xin Tang, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- the First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhaegen PD, Bloemen MC, van der Wal MB, Vloemans AF, Tempelman FR, Beerthuizen GI, van Zuijlen PP. Skin stretching for primary closure of acute burn wounds. Burns. 2014 Dec;40(8):1727-37. doi: 10.1016/j.burns.2014.03.014. Epub 2014 Apr 16. PMID 24746282
- [Background] Verhaegen PDHM, van Trier AJM, Jongen SJM, Vlig M, Nieuwenhuis MK, Middelkoop E, van Zuijlen PPM. Efficacy of skin stretching for burn scar excision: a multicenter randomized controlled trial. Plast Reconstr Surg. 2011 May;127(5):1958-1966. doi: 10.1097/PRS.0b013e31820cf4be. PMID 21228739